CLINICAL TRIAL: NCT07076719
Title: Cell-free DNA Analysis of Spent Embryo Culture Media as a Non-invasive Approach for Preimplantation Genetic Diagnosis
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Collaborators: Assisted Reproductive Technology Unit Life Zena Center, Baghdad, Baghdad Governorate, Iraq (Unknown)
Responsible Party: Principal Investigator, Hatem Awaga, Assistant Professor of Obstetrics and Gynecology, Sohag University
Other Study IDs: CSRE-16-24
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: to Evaluate the Feasibility and Accuracy of Using cfDNA Analysis of Spent Embryo Culture Media as a Non-invasive Approach for PGD
Keywords: Cell-free DNA Analysis; Embryo Culture Media; Preimplantation Genetic Diagnosis
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Paired samples were obtained from 50 embryos that had reached the Day-5 blastocyst stage. From each embryo, we collected the SCM in which it was developing. Subsequently, a corresponding biopsy of the TE was performed and the tissue was collected. All embryos were sourced from a cohort of 20 patients.
  * SCM was harvested after embryo culture with care taken not to include cellular material.
  * TE biopsies were performed according to standard protocols under strict aseptic conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients underwent controlled ovarian stimulation using either:
  o A long down-regulation protocol with buserelin nasal spray (Suprecur, Hoechst, Germany).
  A short protocol incorporating a gonadotropin-releasing hormone (GnRH) antagonist.
  * Gonadotropin Administration: Daily administration included highly purified human menopausal gonadotropin or recombinant FSH. Doses ranged from 150 to 450 IU.
  * Ovulation Trigger: Ovulation was triggered when at least three follicles reached ≥18 mm in diameter. The trigger agents used were either 5,000 IU of hCG or 0.2 mg triptorelin).
  * Oocyte Retrieval: Transvaginal oocyte retrieval was performed 36 hours post-trigger, followed by intracytoplasmic sperm injection (ICSI).
    3. Fertilization and Embryo Culture 4. Trophectoderm (TE) Biopsy 5. Sample Collection and Processing
  Interventions: Diagnostic Test: Trophectoderm (TE) Biopsy; Diagnostic Test: Non-invasive Preimplantation Genetic Diagnosis

INTERVENTIONS:
Diagnostic Test: Trophectoderm (TE) Biopsy — * Blastocyst Grading: Blastocyst grading was based on criteria that classified embryos as good, fair, or poor using the simplified SART embryo scoring system (Heitmann et al., 2013):
    * Good: AA or AB.
    * Fair: BA, BB, BC.
    * Poor: CB or CC.
  * Biopsy Criteria: TE biopsy was performed when an embryo had at least one grade B or better for either the ICM or TE on day 5 of development. When no good-quality blastocysts were available in the same cohort, CC grade blastocysts were biopsied.
  * Biopsy Procedure: 5-8 cells were laser-biopsied from the TE. These cells were then rinsed and tubed for PGT.
  * Cryopreservation: The biopsied embryo was cryopreserved by vitrification (Ref. 90133, Vit Kit-Freeze, Irvine Scientific, Santa Ana, USA) (Richardson et al., 2015).
Diagnostic Test: Non-invasive Preimplantation Genetic Diagnosis — * DNA Contamination Minimization:
    o SCM was harvested after embryo culture with care taken not to include cellular material.
  * Sample Storage:
  * Processing for Genetic Analysis:
    6. DNA Extraction and Sample Preparation 7. Microarray Comparative Genomic Hybridization (aCGH)
  * Chromosomal Assessment:
  * BAC-chip Slides:
  * Labeling and Hybridization:
  * Scanning and Data Acquisition:
  * Data Processing and Analysis:
    8. Validation and Quality Control
  * Robust quality control measures included:

SUMMARY:
This study aims to evaluate the feasibility and accuracy of using cfDNA analysis of spent embryo culture media as a non-invasive approach for PGD. Specifically, the objectives of the study are:

1. To collect SCM from blastocysts of good quality obtained from IVF cycles.
2. To extract cfDNA from the collected SCM using a commercially available kit.
3. To assess the chromosomal content in both cfDNA and gDNA samples via array-based comparative genomic hybridization (aCGH).
4. To compare the results obtained using cfDNA analysis to those obtained using conventional invasive PGD methods, such as blastomere biopsy.
5. To evaluate the potential advantages of using cfDNA analysis of spent embryo culture media for PGD, including reduced risk of harm to the embryo, reduced cost, and increased efficiency.

DETAILED DESCRIPTION:
Materials and Methods:

1. Study Design

   * Type of Study: This is a retrospective study.
   * Location: The study was conducted at the Assisted Reproductive Technology Unit Life Zena Center, Baghdad, Baghdad Governorate, Iraq.
   * Duration: The study was conducted from October 2023 to August 2024.
   * Patient Criteria:

     * Included: All patients referred for PGT-A.
     * Excluded: Patients who had no blastocyst for biopsy were excluded.
   * Ethical Approval: The study was approved by the Committee for the Scientific Research Ethics of Sohag University (CSRE-16-24).
2. Ovarian Stimulation and Oocyte Retrieval

   • Protocols: Patients underwent controlled ovarian stimulation using either:

   o A long down-regulation protocol with buserelin nasal spray (Suprecur, Hoechst, Germany) (Ravhon et al., 2000).

   A short protocol incorporating a gonadotropin-releasing hormone (GnRH) antagonist (Cetrotide, Merck Serono, Germany) (Hohmann et al., 2003).
   * Gonadotropin Administration: Daily administration included highly purified human menopausal gonadotropin (Menopur, Ferring, USA) or recombinant FSH (rFSH; Gonal-F, Serono, Switzerland, or Puregon, MSD, USA). Doses ranged from 150 to 450 IU (Bosch et al., 2024).
   * Ovulation Trigger: Ovulation was triggered when at least three follicles reached ≥18 mm in diameter. The trigger agents used were either 5,000 IU of hCG (Pregnyl, MSD, USA) or 0.2 mg triptorelin (Decapeptyl, Ferring, Sweden) (Schachter et al., 2008)).
   * Oocyte Retrieval: Transvaginal oocyte retrieval was performed 36 hours post-trigger, followed by intracytoplasmic sperm injection (ICSI).
3. Fertilization and Embryo Culture

   * Oocyte Preparation: Collected oocytes were denuded using hyaluronidase (Ref. 10017, Vitrolife, Goteborg, Sweden). They were then incubated for a minimum of one hour before insemination.
   * Insemination: Oocytes were inseminated via ICSI after 4-6 hours of recovery.
   * Initial Culture: Fertilized oocytes were cultured in G-1 medium (Ref. 10127, Vitrolife, Goteborg, Sweden) supplemented with 10% serum substitute supplement (SSS; Ref. 99193, Irvine Scientific, USA).
   * Day 3 Processing: On day 3 of development, each embryo was gently washed and rinsed using a 200 µm pipette (K-FPIP-1170-10, Cook Medical, USA). A ~10 µm hole was drilled in the zona pellucida using a non-contact laser (Saturn 5 Active Laser System, Research Instrument, UK) (Desai et al., 2020).
   * Blastocyst Culture: Embryos were then cultured individually to the blastocyst stage in G-2 medium (Ref. 10131, Vitrolife, Goteborg, Sweden) with 10% SSS.
   * Culture Conditions: The sequential culture was carried out in 30 µl microdrops of media under oil (Ref. 10029, Vitrolife, Goteborg, Sweden). Incubation was performed at 37.0°C in a gas environment of 5% CO₂ and 5% O₂ balanced with N₂ (Zeng et al., 2024).
4. Trophectoderm (TE) Biopsy

   * Blastocyst Grading: Blastocyst grading was based on criteria that classified embryos as good, fair, or poor using the simplified SART embryo scoring system (Heitmann et al., 2013):

     * Good: AA or AB.
     * Fair: BA, BB, BC.
     * Poor: CB or CC.
   * Biopsy Criteria: TE biopsy was performed when an embryo had at least one grade B or better for either the ICM or TE on day 5 of development. When no good-quality blastocysts were available in the same cohort, CC grade blastocysts were biopsied.
   * Biopsy Procedure: 5-8 cells were laser-biopsied from the TE. These cells were then rinsed and tubed for PGT.
   * Cryopreservation: The biopsied embryo was cryopreserved by vitrification (Ref. 90133, Vit Kit-Freeze, Irvine Scientific, Santa Ana, USA) (Richardson et al., 2015).
5. Sample Collection and Processing

   * DNA Contamination Minimization:

     * Embryos and culture media were managed under stringent sterile conditions.
     * Laboratory personnel received comprehensive training in embryo handling protocols and consistently utilized personal protective equipment (masks, caps, gloves).
     * All laboratory materials and equipment were exclusively dedicated to the study to prevent cross-contamination.
     * Meticulous removal of surrounding cumulus cells was performed prior to microinjection in ICSI cycles or at the time of fertilization in conventional IVF cycles to reduce maternal DNA contamination.
     * These practices align with established guidelines for good laboratory practices in IVF settings (Krasic et al., 2021).
   * Sample Collection: Paired samples were obtained from 50 embryos that had reached the Day-5 blastocyst stage. From each embryo, we collected the SCM in which it was developing. Subsequently, a corresponding biopsy of the TE was performed and the tissue was collected. All embryos were sourced from a cohort of 20 patients.

     * SCM was harvested after embryo culture with care taken not to include cellular material.
     * TE biopsies were performed according to standard protocols under strict aseptic conditions.
   * Sample Storage: Samples were stored immediately at -80°C until further processing to prevent degradation of DNA.
   * Processing for Genetic Analysis: TE samples were processed directly for genetic analysis (Magli et al., 2008).
6. DNA Extraction and Sample Preparation

   * cfDNA Extraction: cfDNA was extracted from SCM using the QIAamp Circulating Nucleic Acid Kit (Qiagen, Hilden, Germany). This kit includes a centrifugation step, protein digestion, and silica membrane-based DNA binding optimized for low-yield samples.
   * gDNA Extraction: Genomic DNA (gDNA) was concurrently isolated from the TE biopsy samples using the DNeasy Blood and Tissue Kit (Qiagen), following the manufacturer's instructions (Rubio et al., 2020).
7. Microarray Comparative Genomic Hybridization (aCGH)

   * Chromosomal Assessment: Chromosomal content was assessed in both cfDNA and gDNA samples via array-based comparative genomic hybridization (aCGH).
   * BAC-chip Slides: MACArray Karyo 1440 BAC-chip slides were employed to enable high-resolution, whole-genome profiling.
   * Labeling and Hybridization:

     * Extracted DNA was fluorescently labeled: cfDNA with Cy3 (green) and TE DNA with Cy5 (red).
     * Labeled DNA was hybridized onto oligonucleotide microarrays containing probes across all 23 chromosomes (Mertzanidou et al., 2013).
   * Scanning and Data Acquisition:

     * Post-hybridization, arrays were scanned using an Agilent SureScan microarray scanner (Agilent Technologies, Santa Clara, USA).
     * Signal intensities were quantified, and log₂ ratios of Cy3 to Cy5 fluorescence were calculated to identify chromosomal gains and losses.
   * Data Processing and Analysis:

     * Chromosomal imbalances were analyzed using Agilent CytoGenomics and Genomic Workbench v7.0.4.0 software.
     * Signal data were converted into log₁₀ ratios to determine DNA copy number variations (CNVs).
     * Statistical thresholds were applied to minimize false positives and negatives, regarding established concordance frameworks (Yatsenko et al., 2009).
8. Validation and Quality Control

   • Robust quality control measures included:
   * Negative controls during DNA extraction to detect contamination.
   * Evaluation of hybridization efficiency via reference DNA consistency.
   * Exclusion of results with poor signal-to-noise ratios (Rubio et al., 2019).
9. Statistical Analysis

   * Comparison of Profiles: Chromosomal profiles of cfDNA and TE samples were compared using Chi-square tests.
   * Statistical Significance: P-values <0.05 were considered statistically significant.
10. Software Tools

    * Statistical Analyses: All statistical analyses were performed using SPSS.
    * Visual Data Representations: Visual data representations were generated using GraphPad Prism.

ELIGIBILITY:
Inclusion Criteria:

All patients referred for PGT-A.

Exclusion Criteria:

Patients who had no blastocyst for biopsy were excluded

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — only infertile females who are subjected to ICSI and PGD are eligible for the study
Study Population: Patients underwent controlled ovarian stimulation using either:
  * Gonadotropin Administration:
  * Ovulation Trigger:
  * Oocyte Retrieval:
  * Oocyte Preparation
  * Insemination:
  * Initial Culture
  * Day 3 Processing:
  * Blastocyst Culture:
  * Culture Conditions:
  Trophectoderm (TE) Biopsy Sample Collection and Processing DNA Extraction and Sample Preparation 7. Microarray Comparative Genomic Hybridization (aCGH)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 12 moponths
  Accuracy of using cfDNA analysis of spent embryo culture media as a non-invasive approach for PGD in comparison to traditional trophectoderm biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Unit Life Zena Center, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
We haven't decided yet

REFERENCES:
- [Background] Rubio C, Rienzi L, Navarro-Sanchez L, Cimadomo D, Garcia-Pascual CM, Albricci L, Soscia D, Valbuena D, Capalbo A, Ubaldi F, Simon C. Embryonic cell-free DNA versus trophectoderm biopsy for aneuploidy testing: concordance rate and clinical implications. Fertil Steril. 2019 Sep;112(3):510-519. doi: 10.1016/j.fertnstert.2019.04.038. Epub 2019 Jun 11. PMID 31200971
- [Background] Yatsenko SA, Shaw CA, Ou Z, Pursley AN, Patel A, Bi W, Cheung SW, Lupski JR, Chinault AC, Beaudet AL. Microarray-based comparative genomic hybridization using sex-matched reference DNA provides greater sensitivity for detection of sex chromosome imbalances than array-comparative genomic hybridization with sex-mismatched reference DNA. J Mol Diagn. 2009 May;11(3):226-37. doi: 10.2353/jmoldx.2009.080064. Epub 2009 Mar 26. PMID 19324990
- [Background] Mertzanidou A, Wilton L, Cheng J, Spits C, Vanneste E, Moreau Y, Vermeesch JR, Sermon K. Microarray analysis reveals abnormal chromosomal complements in over 70% of 14 normally developing human embryos. Hum Reprod. 2013 Jan;28(1):256-64. doi: 10.1093/humrep/des362. Epub 2012 Oct 9. PMID 23054067
- [Background] Rubio C, Navarro-Sanchez L, Garcia-Pascual CM, Ocali O, Cimadomo D, Venier W, Barroso G, Kopcow L, Bahceci M, Kulmann MIR, Lopez L, De la Fuente E, Navarro R, Valbuena D, Sakkas D, Rienzi L, Simon C. Multicenter prospective study of concordance between embryonic cell-free DNA and trophectoderm biopsies from 1301 human blastocysts. Am J Obstet Gynecol. 2020 Nov;223(5):751.e1-751.e13. doi: 10.1016/j.ajog.2020.04.035. Epub 2020 May 26. PMID 32470458
- [Background] Magli MC, Van den Abbeel E, Lundin K, Royere D, Van der Elst J, Gianaroli L; Committee of the Special Interest Group on Embryology. Revised guidelines for good practice in IVF laboratories. Hum Reprod. 2008 Jun;23(6):1253-62. doi: 10.1093/humrep/den068. Epub 2008 Mar 28. PMID 18375408
- [Background] Krasic J, Abramovic I, Vrtaric A, Nikolac Gabaj N, Kralik-Oguic S, Katusic Bojanac A, Jezek D, Sincic N. Impact of Preanalytical and Analytical Methods on Cell-Free DNA Diagnostics. Front Cell Dev Biol. 2021 Sep 6;9:686149. doi: 10.3389/fcell.2021.686149. eCollection 2021. PMID 34552921
- [Background] Zeng W, Xiao D, Chen R, Lu Y, Liang W, Sun H. A novel method for gas mixing and distribution in multi-chamber embryo incubators. Technol Health Care. 2024;32(S1):169-181. doi: 10.3233/THC-248015. PMID 38759047
- [Background] Schachter M, Friedler S, Ron-El R, Zimmerman AL, Strassburger D, Bern O, Raziel A. Can pregnancy rate be improved in gonadotropin-releasing hormone (GnRH) antagonist cycles by administering GnRH agonist before oocyte retrieval? A prospective, randomized study. Fertil Steril. 2008 Oct;90(4):1087-93. doi: 10.1016/j.fertnstert.2007.07.1316. Epub 2007 Nov 26. PMID 18023439
- [Background] Bosch E, Alama P, Romero JL, Mari M, Labarta E, Pellicer A. Serum progesterone is lower in ovarian stimulation with highly purified HMG compared to recombinant FSH owing to a different regulation of follicular steroidogenesis: a randomized controlled trial. Hum Reprod. 2024 Feb 1;39(2):393-402. doi: 10.1093/humrep/dead251. PMID 38037188
- [Background] Ravhon A, Aurell R, Lawrie H, Margara R, Winston RM. The significance of delayed suppression using buserelin acetate and recombinant follicle-stimulating hormone in a long protocol in vitro fertilization program. Fertil Steril. 2000 Feb;73(2):325-9. doi: 10.1016/s0015-0282(99)00521-x. PMID 10685537
- [Background] Yu, Y., Liang, X., Wang, W., et al. (2017). Whole-genome sequencing reveals multiple genetic alterations in mesonephric-like adenocarcinomas of the female genital tract. Gynecologic Oncology, 147(3), 617-625.
- [Background] Xiong, B., Ma, H., Zhang, F., Li, Y., Zhou, C., Huang, L., Zhang, Y., Li, R., Wei, J., Liu, P., Wang, J., Tang, F., Liu, Z., Gao, F., & Li, J. (2012). A comparison of human embryo genome-wide copy number profiles was obtained using two different microarray platforms. Reproductive BioMedicine Online, 25(2), 155-161.
- [Background] Wong CC, Loewke KE, Bossert NL, Behr B, De Jonge CJ, Baer TM, Reijo Pera RA. Non-invasive imaging of human embryos before embryonic genome activation predicts development to the blastocyst stage. Nat Biotechnol. 2010 Oct;28(10):1115-21. doi: 10.1038/nbt.1686. Epub 2010 Oct 3. PMID 20890283
- [Background] Wang, Y., Cheng, Q., Meng, L., et al. (2017). Non-invasive detection of genome-wide somatic copy number alterations by liquid biopsies in patients with hepatocellular carcinoma. Oncotarget, 8(33), 54707.
- [Background] Wang, Y., Chen, Y., Zhang, J., Liang, X., Xu, J., Wang, W., Zhang, X., Li, J., Jin, L., & Li, Z. (2018). Whole-genome sequencing of human preimplantation embryos reveals genetic abnormalities and embryonic development. Cell Research, 28(10), 973-987.
- [Background] Wang, L., Zhang, J., Duan, J., et al. (2019). Assessment of human embryos by RNA sequencing, whole-exome sequencing, and karyomapping. Molecular Genetics & Genomic Medicine, 7(7), e00715.
- [Background] Verlinsky, Y., Rechitsky, S., Verlinsky, O., et al. (2013). Preimplantation genetic diagnosis using polar bodies and blastomeres of cleavage stage embryos. Molecular and Cellular Endocrinology, 15(6), 334-339.
- [Background] Vassena R, Boue S, Gonzalez-Roca E, Aran B, Auer H, Veiga A, Izpisua Belmonte JC. Waves of early transcriptional activation and pluripotency program initiation during human preimplantation development. Development. 2011 Sep;138(17):3699-709. doi: 10.1242/dev.064741. Epub 2011 Jul 20. PMID 21775417
- [Background] Scott RT Jr, Upham KM, Forman EJ, Hong KH, Scott KL, Taylor D, Tao X, Treff NR. Blastocyst biopsy with comprehensive chromosome screening and fresh embryo transfer significantly increases in vitro fertilization implantation and delivery rates: a randomized controlled trial. Fertil Steril. 2013 Sep;100(3):697-703. doi: 10.1016/j.fertnstert.2013.04.035. Epub 2013 Jun 1. PMID 23731996
- [Background] Scott RT Jr, Upham KM, Forman EJ, Zhao T, Treff NR. Cleavage-stage biopsy significantly impairs human embryonic implantation potential while blastocyst biopsy does not: a randomized and paired clinical trial. Fertil Steril. 2013 Sep;100(3):624-30. doi: 10.1016/j.fertnstert.2013.04.039. Epub 2013 Jun 15. PMID 23773313
- [Background] Parker, M. T., Knopf, C.W., & Sargent, L. (2007). A comparison of three methods for the estimation of DNA concentration and purity in calf thymus and human leukocytes. Analytical Biochemistry, 361(2), 249-251.
- [Background] Mirkovic J, McFarland M, Garcia E, Sholl LM, Lindeman N, MacConaill L, Dong F, Hirsch M, Nucci MR, Quick CM, Crum CP, McCluggage WG, Howitt BE. Targeted Genomic Profiling Reveals Recurrent KRAS Mutations in Mesonephric-like Adenocarcinomas of the Female Genital Tract. Am J Surg Pathol. 2018 Feb;42(2):227-233. doi: 10.1097/PAS.0000000000000958. PMID 28984674
- [Background] Kirkegaard K, Kesmodel US, Hindkjaer JJ, Ingerslev HJ. Time-lapse parameters as predictors of blastocyst development and pregnancy outcome in embryos from good prognosis patients: a prospective cohort study. Hum Reprod. 2013 Oct;28(10):2643-51. doi: 10.1093/humrep/det300. Epub 2013 Jul 30. PMID 23900207
- [Background] Handyside AH, Kontogianni EH, Hardy K, Winston RM. Pregnancies from biopsied human preimplantation embryos sexed by Y-specific DNA amplification. Nature. 1990 Apr 19;344(6268):768-70. doi: 10.1038/344768a0. PMID 2330030
- [Background] Gardner DK, Lane M, Stevens J, Schlenker T, Schoolcraft WB. Blastocyst score affects implantation and pregnancy outcome: towards a single blastocyst transfer. Fertil Steril. 2000 Jun;73(6):1155-8. doi: 10.1016/s0015-0282(00)00518-5. PMID 10856474
- [Background] Fragouli E, Lenzi M, Ross R, Katz-Jaffe M, Schoolcraft WB, Wells D. Comprehensive molecular cytogenetic analysis of the human blastocyst stage. Hum Reprod. 2008 Nov;23(11):2596-608. doi: 10.1093/humrep/den287. Epub 2008 Jul 29. PMID 18664475
- [Background] Fiorentino F, Bono S, Biricik A, Nuccitelli A, Cotroneo E, Cottone G, Kokocinski F, Michel CE, Minasi MG, Greco E. Application of next-generation sequencing technology for comprehensive aneuploidy screening of blastocysts in clinical preimplantation genetic screening cycles. Hum Reprod. 2014 Dec;29(12):2802-13. doi: 10.1093/humrep/deu277. Epub 2014 Oct 21. PMID 25336713
- [Background] Fiorentino F, Biricik A, Bono S, Spizzichino L, Cotroneo E, Cottone G, Kokocinski F, Michel CE. Development and validation of a next-generation sequencing-based protocol for 24-chromosome aneuploidy screening of embryos. Fertil Steril. 2014 May;101(5):1375-82. doi: 10.1016/j.fertnstert.2014.01.051. Epub 2014 Mar 6. PMID 24613537
- [Background] Zhang P, Zucchelli M, Bruce S, Hambiliki F, Stavreus-Evers A, Levkov L, Skottman H, Kerkela E, Kere J, Hovatta O. Transcriptome profiling of human pre-implantation development. PLoS One. 2009 Nov 16;4(11):e7844. doi: 10.1371/journal.pone.0007844. PMID 19924284
- [Background] Chen AA, Tan L, Suraj V, Reijo Pera R, Shen S. Biomarkers identified with time-lapse imaging: discovery, validation, and practical application. Fertil Steril. 2013 Mar 15;99(4):1035-43. doi: 10.1016/j.fertnstert.2013.01.143. PMID 23499001
- [Background] Chan KC, Jiang P, Zheng YW, Liao GJ, Sun H, Wong J, Siu SS, Chan WC, Chan SL, Chan AT, Lai PB, Chiu RW, Lo YM. Cancer genome scanning in plasma: detection of tumor-associated copy number aberrations, single-nucleotide variants, and tumoral heterogeneity by massively parallel sequencing. Clin Chem. 2013 Jan;59(1):211-24. doi: 10.1373/clinchem.2012.196014. Epub 2012 Oct 11. PMID 23065472